CLINICAL TRIAL: NCT01195311
Title: A Phase I, Open-Label, Dose-Escalation Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of INCB024360 in Patients With Advanced Malignancies
Brief Title: A Dose-escalation Study in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-101
Record Dates: First submitted 2010-08-18; First posted 2010-09-06 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors and Hematologic Malignancy
Keywords: Refractory, Advanced malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INCB024360 (Experimental)
  Interventions: Drug: INCB024360

INTERVENTIONS:
Drug: INCB024360 — INCB024360: 25 mg and 100 mg tablets Doses will be escalated in accordance with the dosing schedule.

SUMMARY:
This is an open label, dose escalation study using a 3 + 3 design to determine if INCB024360 (study drug) is safe, well-tolerated and effective in patients with advanced malignancies. Patients will be enrolled and treated in cohorts of three and each observed a minimum of 28 days before the next group is enrolled and may begin to receive study drug. For subject safety, the first subject in each cohort will be administered drug for one week before the next two subjects in the cohort can begin drug administration. Doses will be escalated unless a dose-limiting toxicity (DLT) is observed in one of three subjects.

An expanded cohort of up to 15 patients may be recruited to further explore safety at the 'maximum tolerated dose' or at a lower, pharmacologically active, dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with neoplastic disease refractory to currently available therapies or for which no effective treatment is available
* Subjects with life expectancy of 12 weeks or longer.
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

Exclusion Criteria:

* Subjects who received any anti-cancer medications in the 21 days prior to receiving their first dose of study medication or 6 weeks for mitomycin-C or nitrosoureas.
* Subjects with history of brain metastases or spinal cord compression.
* Subjects who have undergone a bone marrow or solid organ transplant.
* Subjects who have had major surgery within 4 weeks prior to study entry or had minor surgical procedure within 7 days prior to initiating treatment.
* Subjects with a history of any gastrointestinal condition
* Is receiving any compound that is known to be a potent inducer or inhibitor of CYP3A4
* Subjects with an active autoimmune process or is receiving therapy for an autoimmune disease
* Subjects treated with a serotonin reuptake inhibitor within 3 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by adverse events and dose limiting toxicities | Measured from baseline through follow-up period (measured during cycle 1 weekly and bi monthly thereafter)

SECONDARY OUTCOMES:
Tumor assessment as measured by RECIST criteria | Measured from baseline through treatment cessation. (Measured every other cycle and end of study)
Measurement of IDO inhibition in whole blood measured through blood sampling. | Cycle 1, Day 1 and each 28 day subsequent cycle at Day 1
PK analysis | Full PK at Days 1, 8 (trough only), 15 at Cycle 1 and trough at each subsequent cycle at Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (2):
- United States (2):
  - Chicago, Illinois
  - Philadelphia, Pennsylvania